CLINICAL TRIAL: NCT00654485
Title: A 12 Week Randomized, Double-Blind, Force-Titration, Parallel Group, Multi Centre, Phase IIIb Study to Compare the Efficacy of Rosuvastatin With Atorvastatin and Placebo in the Treatment of Non-Diabetic, Non-Atheroscleric, Metabolic Syndrome Subjects With Raised LDL-C and a 10 Year Risk of CHD >10%
Brief Title: COMETS - Compare the Efficacy of Rosuvastatin With Atorvastatin and Placebo in the Treatment of Non-Diabetic, Non-Atheroscleric, Metabolic Syndrome Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4522IL/0069; D3560C00069
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Metabolic Syndrome
Keywords: Cholesterol; hypercholesterolemia; low density lipoproteins; metabolic syndrome; Rosuvastatin
MeSH Terms: conditions — Metabolic Syndrome; Hypercholesterolemia | interventions — Rosuvastatin Calcium; Atorvastatin

ARMS (2):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (Active Comparator): Atorvastatin
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
  Arms: 1
Drug: Atorvastatin
  Other Names: Lipitor
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy of treatment with rosuvastatin with atorvastatin in reducing Low density lipoprotein cholesterol over 6 weeks of treatment in subjects with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Presence of 3 or more coronary heart disease risk factors as defined by the protocol.
* Fasting low density lipoprotein cholesterol level of > 130 mg/dL.
* Documented history of, or high risk of coronary heart disease or other established atherosclerotic disease.
* Not previously taken statins.

Exclusion Criteria:

* The use of lipid lowering drugs or dietary supplements after Visit 1
* Active arterial disease eg Unstable angina, or recent arterial surgery
* Blood lipid levels above the limits defined in the protocol
* Uncontrolled hypertension, hypothyroidism, alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Estimated)
Dates: Start 2002-05; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol levels following treatment in subjects with metabolic syndrome. | At 6 & 12 weeks

SECONDARY OUTCOMES:
Modification of other lipids and lipoproteins | At 6 & 12 weeks
Modification of insulin resistance, inflammatory markers & glucose metabolism | At 6 & 12 weeks
Safety: adverse events & abnormal laboratory markers | At 6 & 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Anton Stalenhoef, Principal Investigator — University Medical Centre, The Netherlands; Russell Esterline, Study Director — AstraZeneca